CLINICAL TRIAL: NCT06314230
Title: Australian Genomics Of Chronic Allograft Dysfunction Study
Acronym: AUSCAD
Status: Recruiting | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Jennifer Li, Nephrologist and Transplant Physician, Western Sydney Local Health District
Other Study IDs: AUSCAD
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Enrolment is allocated time 0 (baseline). At times 0, 1, 3, 6, 12, 18 and 24 months, patients will be asked to provide blood and urine samples. At time 0, 3, 12 and indication biopsies, a core kidney biopsy if this already being performed as part of clinical care. These samples will biobanked and used to answer the primary questions of this study and consent will be obtained for samples to be used in future research in to renal related disorders.
  After 24months, only medical records will be reviewed in the majority of patients, collecting key outcome measures of kidney function, rejection, major complications or allograft failure (resulting in death or return to dialysis). Patients are invited to participate in the extended follow up phase (after 24months)- where patients may choose to submit blood/urine/tissue samples if an indication biopsy performed as part of their clinical care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: Kidney or kidney-pancreas transplant recipients enrolled into the study prospectively. Risk factors recorded, blood/urine/kidney samples analysed and correlated with outcomes.
  Non-interventional, observational in nature.

SUMMARY:
The goal of the Australian Genomics of Chronic Allograft Dysfunction (AUSCAD) study is a single centre (Westmead Hospital), prospective, observational study, which enrols patients at time of kidney (or kidney-transplant) transplant and tracks the post transplant course. The AUSCAD study aims to generate new knowledge and improve outcomes following kidney transplantation. The primary aim is to determine whether important outcomes (including chronic rejection and graft loss) are correlated with patterns of allograft reactivity, gene expression and susceptibility profiles.

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased donor kidney transplant candidate.
* Biological sex: any
* Ages: 18-75 years.
* Subject must be able to understand and provide informed consent.
* Deceased donor individuals where Research Consent has been obtained from the person consenting to organ donation at the time of organ retrieval.
* Identifiable living donors who have received informed consent and have consented to participate in the project.

Exclusion Criteria:

* Presensitization in living donor recipients prior to transplantation, as determined by site-specific standards, OR positive cross match according to site specific technique in cadaveric donor recipients.
* Recipients of multiple organ transplants, with the exception of kidney/pancreas transplants.
* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* High risk populations including pregnant women, children less than 18 years and prisoners will not be included in the study.
* Non English speaking potential participants who do not understand the requirements of the study will not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, kidney transplant recipients who receive a transplant at Westmead Hospital are eligible for enrolment if they meet the above inclusion/exclusion criteria. They patients can receive a kidney transplant from either kidney-only or kidney-pancreas transplant. They may receive a kidney from either living or deceased donor. Participants are formally enrolled after informed consent and if the transplant proceeds. Participants are allowed to withdraw from the study at any time.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-04-26 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Graft failure | Time Frame: At biopsy or during study follow up after biopsy (expected average 60-months)
  Failure of the kidney transplant, resulting in death or return to dialysis
Allograft rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Any rejection (acute or chronic, borderline, T-cell, antibody or mixed rejection) in the kidney transplant
Gene profile | At biopsy - based on collected tissue sample
  Gene expression or variant profiles of participants

SECONDARY OUTCOMES:
Death | At biopsy or during study follow up after biopsy (expected average over 60-months)
  Death from any cause
Major infectious adverse outcomes | Any time (expected average over 12-months)
  Major viral, bacterial or fungal infections
Major malignancy related adverse outcomes | Any time (expected average over 12-months)
  Major cancers - particularly virally driven malignancies, skin cancers
Major cardiovascular adverse outcomes | Any time (expected average over 12-months)
  4-point MACE: CV death, non-fatal MI, non-fatal stroke, UA requiring hospitalization; and cardiometabolic risks (post-transplant diabetes, dyslipidemia, obesity)
Chronic allograft dysfunction | Any time (expected average 60-months)
  Decline in kidney function in the transplant from the baseline, histologically manifest as fibrosis (interstitial fibrosis and tubular atrophy, IFTA)
BK virus associated nephropathy | At biopsy or during study follow up after biopsy (expected average 12-months)
  BK virus associated nephropathy biopsy evidence of positive SV40 stain in tubules
Albuminuria | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on urine albumin to creatinine ratio
Surrogate end-points | At biopsy or during study follow up after biopsy (expected average 12-months)
  eGFR slow and iBOX score
Delayed graft function (DGF) | At biopsy or during study follow up after biopsy (within 7 days of transplantation)
  Need for dialysis within 7 days of transplantation
Death censored graft loss (DCGL) | At biopsy or during study follow up after biopsy (expected average 12-months)
  Graft loss - excluding cases of death with functioning graft
Treatment resistant rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Persistent rejection despite additional glucocorticoids and/or upscaling of maintenance immunosuppression

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Westmead Institute for Medical Research, Westmead, New South Wales

IPD SHARING:
Plan to Share IPD: No